CLINICAL TRIAL: NCT04512573
Title: Patient Outcomes: Real World Evidence in Rheumatoid Arthritis (POWER)
Status: Completed | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: RA-100-POWER
Record Dates: First submitted 2020-08-05; First posted 2020-08-13 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2023-08

CONDITIONS: Patient Outcomes: Real World Evidence in Rheumatoid Arthritis (POWER)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, real-world observational study in which patients with RA who are initiating treatment with a JAK inhibitor medication will self-report disease activity and treatment satisfaction measures using their own web-enabled device such as a smartphone. Secondary objectives include analyzing the epidemiology and natural history of the disease, its comorbidities, and current treatment practices.

DETAILED DESCRIPTION:
The primary objective of this study is to analyze self-reported disease activity outcomes and treatment satisfaction measures in the real world using a bring-your-own-device approach for patients with rheumatoid arthritis who are initiating a JAKi medication. An exploratory objective is to assess the feasibility of using smartphone or web-based data collection to expand upon the insights gained through the Corrona RA Registry which uses a traditional site-based approach.

POWER is a prospective, non-interventional study that will collect structured real-world data from patients with RA using a patient-centered mobile health application called ArthritisPower™. Patients planning to start treatment with a JAKi medication will self-report disease activity and treatment satisfaction through their first 3 months of therapy using their own web-enabled device such as a smartphone or computer.

Patients will be recruited from the Corrona RA Registry at the time of a routine clinical encounter.

After POWER registration, the remainder of the study is carried out using an automated data collection schedule via the web-based ArthritisPower™ application. Patients may complete assessments using a web browser or by downloading the free ArthritisPower™ application to a smartphone or tablet.

ELIGIBILITY:
Inclusion Criteria:

A patient MUST satisfy all of the following criteria to be eligible for enrollment into the POWER study:

1. Patient is currently participating in the Corrona RA Registry OR is eligible to participate and enrolls into the RA Registry prior to POWER study registration.
2. Patient is willing and able to complete online weekly surveys about their RA using their own computer, tablet,or smartphone and have a valid email address.
3. Patient is literate in English.
4. Patients provides consent for their data to be included in ArthritisPower™ registry in addition to providing consent to participate in the POWER study itself.
5. In conjunction with POWER registration:

   1. A Corrona RA Registry Enrollment or Follow-up visit is conducted (includes both the Provider and Subject questionnaires and most recent Lab/Imaging Results if available)
   2. Patient is newly prescribed* or receives their first dose of one of the following JAK-inhibitor medications: OLUMIANT® (baricitinib), RINVOQ™ (upadacitinib), or XELJANZ / XELJANZ XR® (tofacitinib)**, or any other JAK inhibitor approved during the study period.

      * The decision to treat with a new therapy must precede the decision to recruit the patient into this study. Prior use of a JAK-inhibitor medication does not exclude a patient from enrollment.

        * Patients switching to and from either formula of tofacitinib (Xeljanz 5 mg BID or the "once daily" XR 11 mg version) do not qualify for the POWER study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The following eligibility criteria are designed to select patients for whom study assessments are deemed appropriate. Patients must have attained at least the locally recognized age of consent and provide written or electronic informed consent to participate
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Patterns, effectiveness, and safety of JAK inhibitors currently used in the management of RA | Through Study completion, an average of 10 years
  To analyze self-reported disease activity and treatment satisfaction for patients with RA in the real world at the time of initiation with a JAK inhibitor medication.

SECONDARY OUTCOMES:
Patient Reported: Duration Morning Joint Stiffness | every 6 months for 10 years
Patient Reported: Routine Assessment of Patient Index Data 3 (RAPID3) | every 6 months for 10 years
Patient Reported: PROMIS® Item Bank v.1.0 - Fatigue - Short Form 7a | every 6 months for 10 years
Patient Reported: Compliance Questionnaire for Rheumatology (5-item) | every 6 months for 10 years
Patient Reported: Treatment Satisfaction Questionnaire for Medication (9-item) | every 6 months for 10 years
Patient Reported: PROMIS Anxiety | every 6 months for 10 years
Patient Reported: PROMIS Depression | every 6 months for 10 years
Patient Reported: PROMIS Emotional Support | every 6 months for 10 years
Patient Reported: PROMIS Pain Intensity | every 6 months for 10 years
Patient Reported: PROMIS Pain Interference | every 6 months for 10 years
Patient Reported: PROMIS Physical Function | every 6 months for 10 years
Patient Reported: PROMIS Sleep Disturbance | every 6 months for 10 years)
Patient Reported: PROMIS Satisfaction with Participation in Discretionary Social Activities (Time Frame: every 6 months for 10 years) | every 6 months for 10 years
Patient Reported: PROMIS Ability to Participate in Social Roles and Activities | every 6 months for 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Corrona, LLC, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No